CLINICAL TRIAL: NCT02582788
Title: Bathing Additives in Management of Pediatric Atopic Dermatitis
Brief Title: Bathing Additives in Pediatric Atopic Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Megha M. Tollefson, M.D., Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-003161
Record Dates: First submitted 2015-09-21; First posted 2015-10-21 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bleach (Active Comparator): Patients will use bleach added to their baths twice a week.
  Interventions: Other: Bathing Additive
- Vinegar (Active Comparator): Patients will use vinegar (dilute acetic acid) added to their baths twice a week.
  Interventions: Other: Bathing Additive

INTERVENTIONS:
Other: Bathing Additive

SUMMARY:
The current clinical guidelines for management of atopic dermatitis now recommend bleach baths. This requires simply the addition of regular household bleach to twice-weekly baths. At the Mayo Clinic, dilute acetic acid (vinegar) has been recommended for decades in wet wraps to treat patients hospitalized for their atopic dermatitis. However, this practice has not been widely adopted in the pediatric dermatology community. Will the use of dilute acetic acid (vinegar) in twice weekly baths help manage atopic dermatitis in pediatric patients as well as, or better than, the current accepted guidelines?

ELIGIBILITY:
Inclusion Criteria:

1. Patients from 6 months to 17 years of age
2. Currently residing in US.
3. Follow up visits at 1 month, 3 months and 6 months after initiation of treatment in study (Figure 1).
4. Last follow-up at 1 year in clinic or via written mailed-out survey.
5. Diagnosis of atopic dermatitis AND

   1. Have active signs of bacterial skin infection OR
   2. Any documented suspected history of bacterial skin infection (weeping, crusting, and/or pustules on exam), OR
   3. Prescription for oral antibiotics for skin infection in the past 6 months from any provider). OR
   4. Have been prescribed bleach baths as part of an atopic dermatitis skin care regimen.

Exclusion Criteria:

1. Superficial skin infection without diagnosis of atopic dermatitis
2. Lack of in-clinic follow up assessment at 6 months

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
EASI score at 6 months | 6 months

SECONDARY OUTCOMES:
Courses of antibiotics required | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Megha Tollefson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States